CLINICAL TRIAL: NCT02774005
Title: External Natural History Controlled, Open-Label Intervention Study to Assess the Efficacy and Safety of Long-Term Treatment With Raxone® in Leber's Hereditary Optic Neuropathy (LHON)
Brief Title: Study to Assess the Efficacy and Safety of Raxone in LHON Patients
Acronym: LEROS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNT-IV-005
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Leber's Hereditary Optic Neuropathy (LHON)
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — idebenone

ARMS (1):
- Raxone (Experimental)
  Interventions: Drug: Idebenone

INTERVENTIONS:
Drug: Idebenone
  Other Names: Raxone

SUMMARY:
LEROS is an open-label interventional Phase IV study, designed to further assess the efficacy and safety of Raxone® in the long-term treatment of LHON patients.

ELIGIBILITY:
Inclusion Criteria:

1. Impaired visual acuity in affected eyes due to LHON
2. No explanation for visual loss besides LHON
3. Age more or equal 12 years
4. Onset of symptoms ≤5 years of Baseline
5. Confirmation of either G11778A, G3460A or T14484C LHON mtDNA (for the Intent-to Treat (ITT) population, not required for enrolment)
6. Written informed consent obtained from the patient
7. Ability and willingness to comply with study procedures and visits
8. Women of Childbearing Potential (WCBP) who have a negative urine or serum pregnancy test at Baseline visit and who are willing to use a highly effective contraceptive measure and maintain it until treatment discontinuation.

Exclusion Criteria:

1. Patient has provided natural history data to the Case Record Survey (SNT-CRS-002)
2. Any previous use of idebenone
3. Any other cause of visual impairment (e.g. glaucoma, diabetic retinopathy, AIDS related visual impairment, cataract, macular degeneration, etc.) or any active ocular disorder (uveitis, infections, inflammatory retinal disease, thyroid eye disease, etc.)
4. Known history of clinically significant elevations (greater than 3 times the upper limit of normal) of aspartate aminotransferase (AST), alanine transaminase (ALT) or creatinine
5. Patient has a condition or is in a situation which, in an investigator's opinion may put the patient at significant risk, may confound study results or may interfere significantly with the patient's participation in the study
6. Participation in another clinical trial of any investigational drug within 3 months prior to Baseline
7. Hypersensitivity to the active substance or to any of the following excipients (as listed in section 6.1 of Raxone SmPC): Lactose monohydrate, Microcrystalline cellulose, Croscarmellose sodium, Povidone K25, Magnesium stearate, Colloidal silica, Macrogol 3350, Poly(vinyl alcohol), Talc, Titanium dioxide, Sunset yellow FCF (E110).
8. Women who are pregnant or have a positive pregnancy test at Baseline visit
9. Women who are breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-05; Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (9):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Palo Alto Medical Foundation, Palo Alto, California
  - Stanford Byers Eye Institute, Stanford, California
  - University of Colorado Health Eye Center, Aurora, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Bethesda Neurology, LLC, Bethesda, Maryland
  - Washington University, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - University of Virginia, Charlottesville, Virginia
- AKH - Medizinische Universitaet Wien, Vienna, Austria
- Belgium (4):
  - CHU Saint-Pierre, Brussels
  - Cliniques Universitaire Saint-Luc, Brussels
  - UZ Leuven - Campus Sint-Rafaël, Leuven
  - C. H. U. Sart Tilman, Liège
- UMHAT "Alexandrovska" EAD, Sofia, Bulgaria
- Friedrich-Baur-Institut, München, Germany
- Università di Bologna-Clinica Neurologica-Dipartimento di Scienze Neurologiche, Bologna, Italy
- Poland (5):
  - SPZOZ Spital Uniwersytecki w Krakowie, Oddzial Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM w Szczecinie, Szczecin
  - Samodzielny Publiczny Kliniczny Szpital Okulistyczny, Warsaw
  - Uniwersytecki Szpital Kliniczny, Wroclaw
- Centro Hospitalar de São João, EPE, Porto, Portugal
- Spain (2):
  - Institut Catala de Retina, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
- United Kingdom (4):
  - University Hospital of Wales, Cardiff
  - Moorfields Eye Hospital, London
  - Manchester Royal Eye Hospital, Manchester
  - Queen's Hospital, Romford

REFERENCES:
- [Derived] Yu-Wai-Man P, Carelli V, Newman NJ, Silva MJ, Linden A, Van Stavern G, Szaflik JP, Banik R, Lubinski W, Pemp B, Liao YJ, Subramanian PS, Misiuk-Hojlo M, Newman S, Castillo L, Kociecki J, Levin MH, Munoz-Negrete FJ, Yagan A, Cherninkova S, Katz D, Meunier A, Votruba M, Korwin M, Dziedziak J, Jurkute N, Harvey JP, La Morgia C, Priglinger C, Lloria X, Tomasso L, Klopstock T; LEROS Study Group. Therapeutic benefit of idebenone in patients with Leber hereditary optic neuropathy: The LEROS nonrandomized controlled trial. Cell Rep Med. 2024 Mar 19;5(3):101437. doi: 10.1016/j.xcrm.2024.101437. Epub 2024 Feb 29. PMID 38428428

RESULTS

PARTICIPANT FLOW:
Groups:
- Raxone: Raxone® (idebenone) 150 mg film-coated tablets. 900 mg/day (2 x 150 mg taken orally 3 times daily with meals)
Period: Overall Study
Arm/Group | Raxone
Started | 199 (A total of 199 patients were enrolled in the study. 198 received treatment and were included in the Safety Population. There were 196 patients in the Intent-to-Treat (ITT) population. A total of 181 patients were included in the modified Intent-to-Treat (mITT) population.)
Safety Population | 198
Intent-to-Treat (ITT) Population | 196
Modified Intent-to-Treat (mITT) Population | 181
Completed | 138
Not Completed | 61
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 23
Not completed — Lost to Follow-up | 7
Not completed — Genetic diagnosis reveals that a patient does not harbour a LHON-specific mtDNA mutation | 12
Not completed — Due to Covid-19 lockdown V9 was not completed | 1
Not completed — Pt not willing to perform onsite V9,did not withdraw consent,not triggered by Covid19 situation | 1
Not completed — Death | 1
Not completed — Patient unable to return for visits. Sent medication back to site | 1
Not completed — Lack of compliance with study medication | 4
Not completed — subject is enrolling in a different LHON study that excludes use of idebenone | 1
Not completed — another study | 1
Not completed — cardiologist imposed travel restriction | 1

BASELINE CHARACTERISTICS:
Population: A total of 199 patients were enrolled in the study. 198 received treatment and were included in the Safety Population. There were 196 patients in the ITT population. A total of 181 patients were included in the mITT population.
Arm/Group | Raxone
Number analyzed (Participants) | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29
  Between 18 and 65 years | 164
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 54
  More than one race | 0
  Unknown or Not Reported | 131
Region of Enrollment [Number; unit: participants]
  Austria | 9
  Belgium | 15
  United States | 70
  Poland | 39
  Italy | 12
  United Kingdom | 29
  Bulgaria | 5
  Portugal | 4
  Germany | 4
  Spain | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion (Number) of Eyes With Clinically Relevant Recovery of Visual Acuity From Baseline
Description: Proportion (number) of eyes with clinically relevant recovery of visual acuity (VA) from Baseline or in which Baseline VA better than 1.0 logMAR was maintained at Month 12 in patients treated with Raxone® ≤1 year after the onset of symptoms, compared to matching external natural history control group
Time Frame: 12 months
Population: In the Month 12 dataset with eyes ≤ 1 year after the onset of symptoms at Baseline, used in the evaluation of the primary endpoint, there were 80 patients in the LEROS mITT who contributed 142 eyes for the evaluation.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Raxone
Number analyzed (Participants) | 80
Number analyzed (eyes) | 142
eyes | 60
Statistical Analysis 1: Comparison: Raxone; Test type: Superiority; p = 0.0021, Wald Chi-square; Odds Ratio (OR) = 2.286, 95% CI 2-sided [1.352 to 3.884]

2. Secondary Outcome: Components of the Primary Endpoint: Proportion of Eyes With Clinically Relevant Recovery (CRR) of VA From Baseline at Month 12 Compared to Matching External National History (NH) Control Group
Description: CRR is defined as:
  * Improvement from "off-chart" (the equivalent of Counting fingers, Hand motion, Light perception or No light perception) Visual Acuity to at least 1.6 logMAR value, OR
  * Improvement of at least 0.2 logMAR value within "on-chart" Visual Acuity A patient had a CRR if at least one eye had CRR.
  logMAR = Logarithm of the minimum angle of resolution
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Raxone
Number analyzed (Participants) | 80
Number analyzed (eyes) | 142
eyes | 47
Statistical Analysis 1: Comparison: Raxone; Test type: Superiority; p = 0.0873, Waldi-Chi-Square; Odds Ratio (OR) = 1.646, 95% CI 2-sided [0.929 to 2.918]

3. Secondary Outcome: Components of the Primary Endpoint: Proportion of Eyes in Which Baseline Visual Acuity (VA) Better Than 1.0 logMAR Was Maintained at Month 12 (Clinically Relevant Stabilization) Compared to Matching External NH Control Group
Description: For proportion of eyes in which baseline VA better than 1.0 logMAR was maintained at Month 12 (CRS) compared to matching external NH control group only patients having VA < 1.0 at baseline are taking into account.
  Clinically relevant stabilization (CRS) was defined as maintenance of VA <1.0 logMAR in eyes with VA <1.0 logMAR at Baseline.
  A patient had a CRS if at least one eye had CRS.
  logMAR = Logarithm of the minimum angle of resolution
Time Frame: 12 months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Raxone
Number analyzed (Participants) | 22
Number analyzed (eyes) | 31
eyes | 20
Statistical Analysis 1: Comparison: Raxone; Test type: Superiority; p = 0.0005, Waldi-Chi-Square; Odds Ratio (OR) = 7.323, 95% CI 2-sided [2.339 to 25.912]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 24 months
Arm/Group | Raxone
All-Cause Mortality (participants affected / at risk) | 1/198
Serious Adverse Events (participants affected / at risk) | 27/198
Other Adverse Events (participants affected / at risk) | 148/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raxone (N=198)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Total (Cardiac disorders) | 2 (2)
Total (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Total (General disorders) | 2 (2)
Disease Reoccurance (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Total (Immune system disorders) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1)
Total (Infections and infestations) | 8 (8)
Appendicitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Trichomoniasis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Vulvovaginitis (Infections and infestations) | 1 (1)
Total (Injury, poisoning and procedural complications) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Total (Investigations) | 3 (7)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Urobilinogen urine increased (Investigations) | 1 (1)
Total (Metabolism and nutrition disorders) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Total (Nervous system disorders) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Total (Psychiatric disorders) | 5 (10)
Suicide attempt (Psychiatric disorders) | 3 (3)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Psychotic behaviour (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Total (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Total (Skin and subcutaneous tissue disorders) | 1 (2)
Drug reaction with eosinophilia and systemic (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Total (Social circumstances) | 1 (1)
Miscarriage of partner (Social circumstances) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raxone (N=198)
Total (Blood and lymphatic system disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Total (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Total (Congenital, familial and genetic disorders) | 1 (1)
Hereditary optic atrophy (Congenital, familial and genetic disorders) | 1 (1)
Total (Ear and labyrinth disorders) | 6 (6)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 1 (1)
Total (Endocrine disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1)
Total (Eye disorders) | 15 (22)
Blepharitis (Eye disorders) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 5 (5)
Eyelid pain (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 2 (2)
Photophobia (Eye disorders) | 1 (1)
Photopsia (Eye disorders) | 1 (1)
Pupils unequal (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Visual acuity reduced (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 5 (5)
Total (Gastrointestinal disorders) | 64 (133)
Abdominal discomfort (Gastrointestinal disorders) | 3 (4)
Abdominal migraine (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (10)
Abdominal pain upper (Gastrointestinal disorders) | 13 (14)
Constipation (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dental necrosis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 19 (28)
Dyspepsia (Gastrointestinal disorders) | 5 (9)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (10)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1)
Malpositioned teeth (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 15 (20)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 7 (14)
Vomiting (Gastrointestinal disorders) | 6 (7)
Total (General disorders) | 27 (37)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Cyst (General disorders) | 2 (3)
Fatigue (General disorders) | 8 (8)
Influenza like illness (General disorders) | 4 (5)
Malaise (General disorders) | 5 (5)
Medical device pain (General disorders) | 1 (2)
Pain (General disorders) | 4 (4)
Polyp (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (6)
Total (Hepatobiliary disorders) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1)
Total (Immune system disorders) | 4 (7)
Hypersensitivity (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 3 (6)
Total (Infections and infestations) | 68 (127)
Bacterial abdominal infection (Infections and infestations) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 4 (6)
Bronchitis viral (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 2 (2)
Enterobiasis (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 4 (5)
Gastroenteritis viral (Infections and infestations) | 3 (3)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Hepatitis C (Immune system disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 8 (9)
Lower respiratory tract infection (Infections and infestations) | 3 (5)
Nasopharyngitis (Infections and infestations) | 33 (51)
Oral herpes (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 7 (8)
Skin infection (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (7)
Urinary tract infection (Infections and infestations) | 4 (5)
Viral infection (Infections and infestations) | 1 (1)
Total (Injury, poisoning and procedural complications) | 18 (21)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod sting (Infections and infestations) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (2)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Product administration error (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Total (Investigations) | 50 (132)
Alanine aminotransferase increased (Investigations) | 15 (16)
Aspartate aminotransferase increased (Investigations) | 13 (13)
Bacterial test positive (Investigations) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Blood bicarbonate decreased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (4)
Blood cholesterol increased (Investigations) | 4 (4)
Blood creatine phosphokinase (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 14 (15)
Blood creatinine increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 2 (2)
Blood triglycerides increased (Investigations) | 5 (6)
Blood urea decreased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 2 (2)
Eosinophil count increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 9 (9)
Gastric pH decreased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2)
Liver function test increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Lymphocyte count increased (Investigations) | 3 (3)
Mean cell volume increased (Investigations) | 1 (1)
Mean cell volume increased (Investigations) | 2 (2)
Monocyte count decreased (Investigations) | 1 (1)
Monocyte count increased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 4 (4)
Neutrophil count increased (Investigations) | 3 (3)
Protein urine present (Investigations) | 4 (5)
Red blood cell count decreased (Investigations) | 2 (2)
Transaminases increased (Investigations) | 1 (1)
Urinary sediment present (Investigations) | 2 (2)
Urine ketone body present (Investigations) | 2 (2)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3)
White blood cells urine positive (Investigations) | 1 (1)
Total (Metabolism and nutrition disorders) | 6 (10)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Total (Musculoskeletal and connective tissue disorders) | 25 (38)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (13)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Total (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Total (Nervous system disorders) | 49 (152)
Burning sensation (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 37 (131)
Hyperaesthesia (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Ophthalmic migraine (Nervous system disorders) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Total (Psychiatric disorders) | 25 (34)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1)
Anger (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4)
Confusional state (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 8 (8)
Depressive symptom (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Irritability (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Polydipsia psychogenic (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2)
Suicidal behaviour (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Total (Renal and urinary disorders) | 9 (12)
Chromaturia (Renal and urinary disorders) | 3 (6)
Glycosuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Urine abnormality (Psychiatric disorders) | 3 (3)
Total (Reproductive system and breast disorders) | 6 (12)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (9)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Total (Respiratory, thoracic and mediastinal disorders) | 32 (65)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (22)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Total (Social circumstances) | 3 (3)
Orthosis user (Social circumstances) | 1 (1)
Pregnancy of partner (Skin and subcutaneous tissue disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (7)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Total (Vascular disorders) | 6 (6)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The below agreement was included in the Clinical Trial Agreement : Study Team Member agrees not to publish or refer to the study, in whole or in part, without the prior expressed written consent of the sponsor. Study team member will not use the name of the sponsor or [name of the study co-ordinating Contract Research Organization (CRO)] in connection with any publication or promotion without sponsor's or [name co-ordinating CRO]'s prior, written consent.

DOCUMENTS (2):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT02774005/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT02774005/SAP_001.pdf